CLINICAL TRIAL: NCT00945659
Title: Use of Continuous Glucose Sensors by Adolescents With Inadequate Diabetic Control
Acronym: CGM-Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Timothy Wysocki, Principal Research Scientist and Center Director, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01DK080831 (NIH); 1R01DK080831 (NIH)
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Standard of Care; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: 3 group (Standard Care: Continuous Glucose Monitor; Continuous Glucose Monitor + Behavior Therapy) X 4 time points (0, 3, 6, and 9 months) Repeated measures randomized treatments design.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Care (Active Comparator): Standard Care constitutes intensified diabetes management, an enrollment criterion for the study, consisting of either continuous subcutaneous insulin infusion (insulin pump) or multiple daily injections using a "basal-bolus" approach. All patients must be using carbohydrate counting and have prescribed correction factors for targeted insulin bolus dose adjustments.
  Interventions: Other: Standard Care
- Continuous Glucose Sensor (Active Comparator): Patients will have the same diabetes management regimen as those in the Standard Care group. In addition they will be given a continuous glucose sensor, receive expert instruction in its use, and be guided by a physician and diabetes educator in achieving glycemic benefits through retrospective and real-time interpretation of CGS results and by learning to respond judiciously to the various CGS alarms.
  Interventions: Device: Continuous Glucose Sensor
- CGS + Behavior Therapy (Experimental): Patients in the use group will receive the same medical management as the Continuous Glucose Sensor group above. In addition, they will have 6 scheduled encounters with a behavior therapist that are designed to reduce or eliminate typical behavioral and/or psychological barriers to optimal use of CGS as part of diabetes care.
  Interventions: Behavioral: CGS + Behavior Therapy

INTERVENTIONS:
Device: Continuous Glucose Sensor — Education and medical management to promote optimal therapeutic benefit from adding use of a continuous glucose sensor to daily diabetes management.
  Arms: Continuous Glucose Sensor
Other: Standard Care — Intensified diabetes management based on either insulin pump or multiple daily injection insulin regimen, employing carbohydrate counting and a bolus dose correction factor for adjusting insulin doses.
  Arms: Standard Care
Behavioral: CGS + Behavior Therapy — Patients in this group will receive 6 scheduled encounters with a behavior therapist who will assist the adolescent and parent in reducing or eliminating common behavioral and psychological barriers to achieving optimal benefit from CGS use in diabetes care.
  Arms: CGS + Behavior Therapy

SUMMARY:
The incorporation of continuous glucose sensors (CGS) into management of type 1 diabetes in adolescence could improve treatment outcomes. But, behavioral barriers may prevent adolescents from enjoying optimal benefits from this new technology. This study will randomize adolescents (11 to not yet 17 years old) with type 1 diabetes for at least 2 years who are not achieving targeted HbA1c levels (> 7.5%) to continue in standard care (SC), to add continuous glucose monitoring (CGM) to their care with appropriate education and medical management (CGS) or to add CGM to their care as above but to also receive support and assistance from a behavior therapist who will assist the patient and family in optimizing the adolescents' therapeutic benefit from CGS (CGS+BT). A variety of outcomes will be measured, including blood glucose control, quality of life, and CGS satisfaction and impact. An enrollment criterion for this study is that the adolescent must have established consistent care for type 1 diabetes at a Nemours Children's Clinic location either in Wilmington, DE, Philadelphia, PA, Orlando, FL or Pensacola, FL for at least 12 months prior to enrollment in the study. Adolescents treated elsewhere are not eligible to enroll in the study.

DETAILED DESCRIPTION:
Management of type 1 diabetes mellitus (T1DM) in adolescents is very difficult and innovative approaches are needed to help them achieve better glycemic control and behavioral outcomes. Continuous glucose sensors (CGS) have been refined progressively and provide acceptably accurate, nearly continuous estimates of glucose levels and trends. This increased quality and quantity of glucose data could be an excellent adjunct to conventional self-monitoring of blood glucose, permitting more informed diabetes decision-making. CGS could yield medical, educational and psychological benefits for adolescents with T1DM, but those with extremely variable self-management habits and suboptimal glycemic control may not realize these benefits readily. We hypothesize that a targeted, family-focused behavioral intervention could optimize benefit from adding CGS to T1DM therapy for youths with glycosylated hemoglobin (HbA1c) > 7.5%. A multi-site sample of 150 adolescents with T1DM and HbA1C of 7.5% to 10.0% will be randomized to either Standard Care for T1DM (SC), or to augmentation of SC with 9 months' use of a CGS device (CGS) or use of a CGS device supplemented with a targeted behavior therapy intervention (CGS+BT). Multiple measures of glycemic control, glycemic variability and health care use will be obtained during the study and there will be periodic assessments of demographic factors, diabetes self-management, family relations and psychological adjustment. Three specific aims will be addressed: 1. Evaluate whether CGS+BT yields more improvement in glycemic outcomes than CGS or SC; 2. Evaluate whether CGS+BT yields more improvement in behavioral outcomes than CGS or SC; and 3. Identify behavioral variables that mediate and moderate glycemic benefit from use of the CGS device. The study will also compare the cost effectiveness of CGS and CGS+BT relative to SC and evaluate the predictive utility of various indices of glycemic variability in youths. We hypothesize that, compared with SC and CGS, CGS+BT will yield significantly better biomedical outcomes (HbA1C; severe hypoglycemia; glycemic variability; proportion of glucose readings in the normal range) and behavioral outcomes (treatment adherence; parent adolescent teamwork; diabetes-related family conflict; quality of life; fear of hypoglycemia; and treatment satisfaction). After the 9 month randomized trial, all youths will be allowed to use the CGS device during an additional 3-month continuation phase. Statistical analyses will be based on individual growth modeling techniques. The application capitalizes on the Principal Investigator's prior and ongoing funded research on family management of T1DM, including trials of family-focused behavioral interventions, intensive therapy regimens, and clinical evaluations of continuous glucose sensors. The proposed study will determine whether a targeted behavioral intervention improves CGS benefits among adolescents with previously inadequate glycemic control. These results could demonstrate that adolescents with previously suboptimal diabetic control could realize multiple benefits from CGS use if they are provided with a specialized behavioral intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age of adolescent > 11 years and < 17 years. This age range was chosen because families of adolescents often struggle with diabetes management. Youths > 18 years old may be likely to leave home during the study.
2. Diagnosis of type 1 diabetes based on the clinician's best judgment regarding the adolescent's proper diagnostic category.
3. Duration of type 1 diabetes > 2 years or > 1 year with negligible stimulated c-peptide level, to exclude those with significant residual pancreatic insulin production.
4. Treatment of diabetes for the 6 months prior to enrollment must consist of an intensified regimen including either daily use of an insulin pump or 3 or more daily insulin injections with pre-meal insulin doses calculated using a correction factor that considers prevailing blood glucose levels and planned carbohydrate intake.
5. Adolescent must have established diabetes care at a participating Nemours Children's Clinic site as evidenced by at least two diabetes clinic visits within the prior 12 months.
6. Most recent HbA1C > 7.5% and < 10.0% or mean HbA1C over the prior 12 months within that same range.
7. Intention to remain in the same region and to maintain diabetes care at the enrolling center for 12 months.
8. Family has working telephone service.

Exclusion Criteria:

1. Youth has not used a CGM device with real-time glucose feedback for clinical management of diabetes within the prior 6 months. Intermittent or one-time use of "blinded" CGM devices for retrospective analysis only is permissible.
2. Absence of any other medical conditions that, in the opinion of the attending endocrinologist, would impede completion of the study protocol.
3. Youths may not be on daily glucocorticoid medications due to hyperglycemic effects of these agents.
4. Not enrolled in special education for mental retardation, autism or severe behavior disorders.
5. Child not in an inpatient psychiatric unit or day treatment program during the 6 months prior to enrollment.
6. Primary diabetes caregiver not diagnosed or in treatment for major depression, psychosis, bipolar disorder or substance use disorder within the 6 months prior to enrollment; Child not in an inpatient psychiatric unit or day treatment program during the 6 months prior to enrollment.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2009-08; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Wysocki, Ph.D., Principal Investigator — Nemours Children's Clinic Jacksonville
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Started | 39 | 40 | 37
Baseline | 39 | 40 | 37
3-Months | 38 | 39 | 35
6-Months | 31 | 29 | 25
9-Months | 32 | 20 | 20
12-Months | 32 | 20 | 20
Completed | 32 | 20 | 20
Not Completed | 7 | 20 | 17
Not completed — Lost to Follow-up | 7 | 20 | 17

BASELINE CHARACTERISTICS:
Groups:
- CGS + Behavior Therapy: Patients in this group will receive the same medical management as the Continuous Glucose Sensor group above. In addition, they will have 6 scheduled encounters with a behavior therapist that are designed to reduce or eliminate typical behavioral and/or psychological barriers to optimal use of CGS as part of diabetes care.
  CGS + Behavior Therapy: Patients in this group will receive 6 scheduled encounters with a behavior therapist who will assist the adolescent and parent in reducing or eliminating common behavioral and psychological barriers to achieving optimal benefit from CGS use in diabetes care.
- Total: Total of all reporting groups
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy | Total
Number analyzed (Participants) | 38 | 39 | 35 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] — Adolescent Age in Years
  years | 13.61 (1.76) | 13.62 (1.82) | 13.46 (1.98) | 13.56 (1.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 23 | 61
  Male | 19 | 20 | 12 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 5 | 12
  Not Hispanic or Latino | 34 | 34 | 30 | 98
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 3 | 9
  White | 32 | 32 | 28 | 92
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 4 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 39 | 35 | 112
Glycated Hemoglobin Level (%) [Mean (Standard Deviation); unit: Percentage of hemoglobin] — Glycated hemoglobin level expressed as percentage of hemoglobin molecules bound to glucose molecules.
  Percentage of hemoglobin | 8.84 (0.95) | 9.03 (1.07) | 9.24 (0.83) | 9.03 (0.96)

OUTCOME MEASURES:

1. Primary Outcome: Glycated Hemoglobin (HbA1c)
Description: Glycated hemoglobin (HbA1c) expressed as a percentage of hemoglobin molecules bound to glucose.
Time Frame: Baseline, 3, 6, 9 months
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin molecules
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Number analyzed (Participants) | 38 | 39 | 35
percentage of hemoglobin molecules
  Baseline | 8.84 (0.95) | 9.03 (1.07) | 9.24 (0.83)
  3-Months | 9.14 (1.38) | 9.06 (1.10) | 8.96 (0.84)
  6-Months | 8.95 (1.14) | 9.35 (1.30) | 9.09 (1.71)
  9-Months | 8.96 (1.04) | 9.51 (1.37) | 9.05 (1.14)
Statistical Analysis 1: Comparison: Standard Care vs Continuous Glucose Sensor; Test type: Superiority; p = 0.86, Generalized Estimating Equation; Mean Difference (Net) = -.003, 95% CI 2-sided [-0.43 to 0.36], Standard Deviation 0.2
Statistical Analysis 2: Comparison: Standard Care vs CGS + Behavior Therapy; Test type: Superiority; p = 0.03, Generalized Estimating Equation; Mean Difference (Net) = -0.41, 95% CI 2-sided [-0.78 to -0.04], Standard Error of Mean 0.19

2. Secondary Outcome: Diabetes Technology Questionnaire-Adolescents
Description: Adolescent's total score on the DTQ-Current items. Range 30-150. Higher scores indicate more favorable satisfaction with and impact of the package of diabetes technology (e.g. pump, meter, CGM, etc.) in use by the patient during the prior 3 months.
Time Frame: Baseline, 3 6, 9 months
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Number analyzed (Participants) | 38 | 39 | 35
Total score
  Baseline | 96.50 (18.29) | 101.73 (23.26) | 105.16 (27.89)
  3-Months | 102.24 (24.44) | 92.50 (20.28) | 105.95 (27.7)
  6-Months | 109.32 (19.57) | 107.51 (21.65) | 113.19 (24.41)
  9-Months | 112.62 (23.69) | 103.00 (21.95) | 103.93 (27.47)
Statistical Analysis 1: Comparison: Standard Care vs Continuous Glucose Sensor; Test type: Superiority; p = 0.03, Generalized Estimating Equation; Mean Difference (Net) = -10.05, 95% CI 2-sided [-19.30 to -0.81], Standard Deviation 4.72
Statistical Analysis 2: Comparison: Standard Care vs CGS + Behavior Therapy; Test type: Superiority; p = 0.88, Generalized Estimating Equation; Mean Difference (Net) = -0.82, 95% CI 2-sided [-11.54 to 9.9], Standard Deviation 5.47

3. Secondary Outcome: Diabetes Technology Questionnaire-Parents' Total Scores on DTQ Current Items
Description: Parents' ratings of impact and satisfaction with the diabetes devices currently in use (e.g. pump, meter, CGM etc.) Score range from 30-150. Higher score signify greater satisfaction and impact.
Time Frame: Baseline, 3, 6, 9 months
Measure: Mean (Standard Deviation); unit: Total scores
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Number analyzed (Participants) | 38 | 39 | 35
Total scores
  Baseline | 90.06 (17.39) | 91.68 (21.34) | 86.87 (27.01)
  3-Months | 90.48 (25.03) | 93.78 (21.35) | 95.92 (26.76)
  6-Months | 93.21 (25.82) | 94.70 (19.25) | 96.27 (29.64)
  9-Months | 104.65 (21.61) | 96.79 (18.15) | 98.53 (23.31)
Statistical Analysis 1: Comparison: Standard Care vs Continuous Glucose Sensor; Test type: Superiority; p = 0.49, Generalized Estimating Equation; Generalized Estimating Equation = -3.45, 95% CI 2-sided [-13.21 to 6.32], Standard Deviation 4.98
Statistical Analysis 2: Comparison: Standard Care vs CGS + Behavior Therapy; Test type: Superiority; p = 0.66, Generalized Estimating Equation; Mean Difference (Net) = 2.53, Standard Deviation 5.76

4. Secondary Outcome: Blood Glucose Monitoring Communication Questionnaire-Adolescent
Description: Adolescent report of communication with parents about blood glucose monitoring and results. Range 8-24. Higher scores indicate more negative communication about BG results.
Time Frame: Baseline, 3, 6, 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Number analyzed (Participants) | 38 | 39 | 35
units on a scale
  Baseline | 14.24 (2.84) | 14.46 (3.04) | 14.29 (3.5)
  3-Months | 14.46 (2.80) | 14.43 (3.72) | 13.54 (4.21)
  6-Months | 13.76 (3.88) | 14.57 (4.36) | 13.16 (4.27)
  9-months | 14.25 (3.76) | 14.03 (4.49) | 14.47 (4.35)
Statistical Analysis 1: Comparison: Standard Care vs Continuous Glucose Sensor; Test type: Superiority; p = 0.64, Generalized Estimating Equation; Mean Difference (Net) = 0.40, 95% CI 2-sided [-1.29 to 2.08], Standard Deviation 0.86
Statistical Analysis 2: Comparison: Standard Care vs CGS + Behavior Therapy; Test type: Superiority; p = 0.65, Generalized Estimating Equation; Mean Difference (Net) = -0.41, 95% CI 2-sided [-2.22 to 1.39], Standard Deviation 0.92

5. Secondary Outcome: Blood Glucose Monitoring Communication Questionnaire-Parents
Description: Parents perspectives of communication with adolescent around blood glucose monitoring and results. Score range 8-24. Higher scores signify more negative communication about BG results.
Time Frame: Baseline, 3, 6, 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Number analyzed (Participants) | 38 | 39 | 35
units on a scale
  Baseline | 14.08 (2.83) | 14.59 (2.87) | 14.29 (3.50)
  3-Months | 14.46 (3.05) | 15.13 (3.29) | 12.84 (3.36)
  6-Months | 15.16 (3.14) | 15.41 (3.43) | 12.72 (3.92)
  9-Months | 14.46 (3.39) | 14.36 (1.95) | 13.69 (3.57)
Statistical Analysis 1: Comparison: Standard Care vs Continuous Glucose Sensor; Test type: Superiority; p = 0.99, Generalized Estimating Equation; Mean Difference (Net) = 0.71, 95% CI 2-sided [-123.56 to 124.97], Standard Deviation 63.40
Statistical Analysis 2: Comparison: Standard Care vs CGS + Behavior Therapy; Test type: Superiority; p = 0.93, Generalized Estimating Equation; Mean Difference (Net) = -1.22, 95% CI 2-sided [-28.26 to 25.83], Standard Deviation 13.81

6. Secondary Outcome: Diabetes Family Conflict Scale-Adolescent
Description: Adolescent ratings of degree of diabetes-related family conflict. Score range 19-57. Higher scores indicate more frequent family conflict around diabetes.
Time Frame: Baseline, 3, 6, 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Number analyzed (Participants) | 38 | 39 | 35
units on a scale
  Baseline | 27.72 (7.25) | 27.54 (7.92) | 27.59 (8.37)
  3-Months | 27.41 (7.22) | 29.70 (9.57) | 25.26 (8.16)
  6-Months | 27.07 (9.31) | 28.73 (8.48) | 24.35 (7.69)
  9-Months | 26.68 (9.31) | 27.29 (6.56) | 25.06 (9.09)
Statistical Analysis 1: Comparison: Standard Care vs Continuous Glucose Sensor; Test type: Superiority; p = 0.43, Generalized Estimating Equation; Mean Difference (Net) = 1.17, 95% CI 2-sided [-1.70 to 4.04], Standard Deviation 1.47
Statistical Analysis 2: Comparison: Standard Care vs CGS + Behavior Therapy; Test type: Superiority; p = 0.08, Generalized Estimating Equation; Mean Difference (Net) = -2.59, 95% CI 2-sided [-5.50 to 0.32], Standard Deviation 1.87

7. Secondary Outcome: Diabetes Family Conflict Scale-Parent
Description: Parents' ratings of degree of diabetes-related family conflict. Score range 19-57. Higher scores indicate more family conflict around diabetes.
Time Frame: Baseline, 3, 6, 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Number analyzed (Participants) | 38 | 39 | 35
units on a scale
  Baseline | 28.76 (7.27) | 27.76 (5.12) | 27.75 (6.06)
  3-Months | 29.36 (8.48) | 30.29 (7.82) | 24.85 (5.13)
  6-Months | 30.62 (8.68) | 29.05 (8.44) | 24.85 (5.29)
  9-Months | 26.68 (5.38) | 29.43 (6.85) | 24.18 (3.19)
Statistical Analysis 1: Comparison: Standard Care vs Continuous Glucose Sensor; Test type: Superiority; p = 0.43, Generalized Estimating Equation; Mean Difference (Net) = 1.32, 95% CI 2-sided [-1.94 to 4.56], Standard Deviation 1.66
Statistical Analysis 2: Comparison: Standard Care vs CGS + Behavior Therapy; Test type: Superiority; p = .007, Generalized Estimating Equation; Mean Difference (Net) = -3.71, 95% CI 2-sided [-6.38 to -1.04], Standard Deviation 1.36

8. Secondary Outcome: Diabetes Family Responsibility Questionnaire-Adolescent
Description: Adolescent's self-ratings of their degree of responsibility for 38 diabetes tasks. Score range 0-76. Lower scores indicate greater adolescent responsibility for diabetes care.
Time Frame: Baserline, 3, 6, 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Number analyzed (Participants) | 38 | 39 | 35
units on a scale
  Baseline | 31.53 (4.74) | 31.15 (5.04) | 31.38 (5.48)
  3-Months | 31.20 (5.36) | 31.56 (4.15) | 30.48 (5.02)
  6-Months | 29.85 (4.88) | 29.96 (4.15) | 28.71 (5.53)
  9-Months | 29.65 (4.72) | 30.25 (4.16) | 29.56 (5.21)
Statistical Analysis 1: Comparison: Standard Care vs Continuous Glucose Sensor; Test type: Superiority; p = 0.75, Generalized Estimating Equation; Mean Difference (Net) = 0.39, 95% CI 2-sided [-2.02 to 2.79], Standard Deviation 1.23
Statistical Analysis 2: Comparison: Standard Care vs CGS + Behavior Therapy; Test type: Superiority; p = 0.78, Generalized Estimating Equation; Mean Difference (Net) = -0.39, 95% CI 2-sided [-3.09 to 2.32], Standard Deviation 1.38

9. Secondary Outcome: Diabetes Family Responsibility Questionnaire-Parent
Description: Parent ratings of adolescent's degree of responsibility for 38 diabetes tasks. Score range 0-76. Lower scores indicate great adolescent responsibility for diabetes care tasks.
Time Frame: Baseline, 3, 6, 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Number analyzed (Participants) | 38 | 39 | 35
units on a scale
  Baseline | 34.44 (4.05) | 35.19 (5.22) | 33.97 (5.03)
  3-Months | 34.22 (5.31) | 34.23 (6.32) | 33.62 (4.24)
  6-Months | 32.50 (4.19) | 34.35 (6.47) | 32.30 (5.19)
  9-Months | 32.00 (4.01) | 35.10 (5.15) | 33.28 (5.16)
Statistical Analysis 1: Comparison: Standard Care vs Continuous Glucose Sensor; Test type: Superiority; p = 0.58, Generalized Estimating Equation; Mean Difference (Net) = 0.72, 95% CI 2-sided [-1.86 to 3.29], Standard Deviation 1.31
Statistical Analysis 2: Comparison: Standard Care vs CGS + Behavior Therapy; Test type: Superiority; p = 0.41, Generalized Estimating Equation; Mean Difference (Net) = -0.93, 95% CI 2-sided [-3.17 to 1.3], Standard Deviation 1.14

10. Secondary Outcome: Diabetes Self Management Profile-Adolescent
Description: Adolescent self-report of diabetes management behaviors. Score range 0-86. Higher scores indicate more meticulous diabetes treatment adherence.
Time Frame: Baseline, 3, 6, 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Number analyzed (Participants) | 38 | 39 | 35
units on a scale
  Baseline | 57.05 (14.71) | 60.25 (13.68) | 59.38 (12.79)
  3-Months | 56.82 (13.88) | 58.73 (14.19) | 57.79 (13.47)
  6-Months | 59.36 (14.03) | 61.14 (13.22) | 59.07 (13.29)
  9-Months | 55.43 (14.49) | 58.74 (13.74) | 58.13 (14.17)
Statistical Analysis 1: Comparison: Standard Care vs Continuous Glucose Sensor; Test type: Superiority; p = 0.46, Generalized Estimating Equation; Mean Difference (Net) = 1.95, 95% CI 2-sided [-3.26 to 7.15], Standard Deviation 2.66
Statistical Analysis 2: Comparison: Standard Care vs CGS + Behavior Therapy; Test type: Superiority; p = 0.24, Generalized Estimating Equation; Mean Difference (Net) = -3.01, 95% CI 2-sided [-7.99 to 1.96], Standard Deviation 2.54

11. Secondary Outcome: Diabetes Self Management Profile-Parent
Description: Parent report of adolescent's diabetes self-management behaviors. Score range 0-86. Higher scores indicate more meticulous diabetes treatment adherence.
Time Frame: Baseline, 3, 6, 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Number analyzed (Participants) | 38 | 39 | 35
units on a scale
  Baseline | 52.76 (13.81) | 55.45 (14.06) | 55.94 (13.37)
  3-Months | 54.15 (13.49) | 58.18 (14.51) | 59.07 (12.84)
  6-Months | 51.93 (14.17) | 59.26 (14.37) | 60.19 (14.28)
  9-Months | 54.38 (13.65) | 57.16 (13.58) | 58.73 (14.11)
Statistical Analysis 1: Comparison: Standard Care vs Continuous Glucose Sensor; Test type: Superiority; p = 0.93, Generalized Estimating Equation; Mean Difference (Net) = 0.31, 95% CI 2-sided [-6.33 to 6.91], Standard Deviation 3.37
Statistical Analysis 2: Comparison: Standard Care vs CGS + Behavior Therapy; Test type: Superiority; p = 0.45, Generalized Estimating Equation; Mean Difference (Net) = -2.21, 95% CI 2-sided [-8.01 to 3.57], Standard Deviation 2.95

12. Secondary Outcome: Hypoglycemia Fear Survey-Adolescent
Description: Adolescent worry and behavior related to apprehension of low BG episodes. Score range 24-72. Higher scores indicate greater fear and avoidance of hypoglycemia
Time Frame: Baseline, 3, 6, 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Number analyzed (Participants) | 38 | 39 | 35
units on a scale
  Baseline | 36.94 (11.69) | 35.8 (12.46) | 35.39 (12.55)
  3-Months | 35.95 (12.86) | 37.15 (15.34) | 31.00 (12.79)
  6-Months | 34.01 (12.98) | 35.30 (11.55) | 32.19 (16.12)
  9-Months | 27.91 (9.31) | 38.00 (15.38) | 35.24 (14.52)
Statistical Analysis 1: Comparison: Standard Care vs Continuous Glucose Sensor; Test type: Superiority; p = 0.81, Generalized Estimating Equestion; Mean Difference (Net) = -0.77, 95% CI 2-sided [-7.15 to 5.62], Standard Deviation 3.26
Statistical Analysis 2: Comparison: Standard Care vs CGS + Behavior Therapy; Test type: Superiority; p = 0.72, Generalized Estimating Equation; Mean Difference (Net) = 0.99, 95% CI 2-sided [-4.11 to 6.08], Standard Deviation 2.63

13. Secondary Outcome: Hypoglycemia Fear Survey-Parent
Description: Parental worry and behavior related to apprehension of low BG events. Score range 24-72. Higher scores indicate greater parental fear and avoidance of hypoglycemia.
Time Frame: Baseline, 3, 6, 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
Number analyzed (Participants) | 38 | 39 | 35
units on a scale
  Baseline | 43.31 (15.2) | 43.5 (11.52) | 44.09 (13.85)
  3-Months | 40.07 (12.00) | 41.56 (10.72) | 39.79 (9.49)
  6-Months | 45.59 (12.70) | 43.14 (9.49) | 41.76 (16.71)
  9-Months | 38.48 (11.62) | 39.87 (7.48) | 40.67 (11.24)
Statistical Analysis 1: Comparison: Standard Care vs Continuous Glucose Sensor; Test type: Superiority; p = 0.71, Generalized Estimating Equation; Mean Difference (Net) = 0.99, 95% CI 2-sided [-4.11 to 6.08], Standard Deviation 2.6
Statistical Analysis 2: Comparison: Standard Care vs CGS + Behavior Therapy; Test type: Superiority; p = 0.68, Generalized Estimating Equation; Mean Difference (Net) = -1.16, 95% CI 2-sided [-6.74 to 4.43], Standard Deviation 2.85

ADVERSE EVENTS:
Time Frame: 9 months for each participant
Arm/Group | Standard Care | Continuous Glucose Sensor | CGS + Behavior Therapy
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/39 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39 | 0/35
Other Adverse Events (participants affected / at risk) | 0/38 | 0/39 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT00945659/Prot_SAP_000.pdf
  • Informed Consent Form (2012-11-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT00945659/ICF_001.pdf